CLINICAL TRIAL: NCT00662727
Title: Randomized, Placebo Controlled, Double Blind Clinical Trial Evaluating the Treatment of Patients With Refractory Angina Pectoris With Low Intensity Extracorporeal Shockwave Therapy Device
Brief Title: Extracorporeal Shockwave Therapy for the Treatment of Refractory Angina Pectoris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medispec (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESMR-RCT-IL
Record Dates: First submitted 2008-04-14; First posted 2008-04-21 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Refractory Angina Pectoris
Keywords: Extracorporeal Shockwave Therapy; Myocardial Ischemia; Refractory Angina
MeSH Terms: conditions — Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): A - Treatment group. Patients in this group receive actual shockwave therapy.
  Interventions: Device: Cardiac Extracorporeal Shockwave Therapy generator (Cardiospec)
- B (Placebo Comparator): Placebo group. This group of patients undergo the same procedure as the treatment group, however shockwaves are not delivered to the heart.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Cardiac Extracorporeal Shockwave Therapy generator (Cardiospec) — Energy Density - 0.09 mJ/mm2
  Other Names: Cardiospec; ESMR therapy; Extracorporeal Shockwave Myocardial Revascularization
  Arms: A
Device: Placebo — Placebo
  Arms: B

SUMMARY:
Low intensity shockwaves have been proven in animal studies to induce local growth of new blood vessels from existing ones.

The hypothesis of this study is that shockwave therapy could improve the symptoms of patients with refractory angina not amenable to revascularization with angioplasty or bypass surgery.

DETAILED DESCRIPTION:
Low intensity shockwaves (1/10 the ones used in Lithotripsy) are delivered to myocardial ischemic tissue. Shockwaves are created by a special generator and are focused using a shockwave applicator device. The treatment is guided by standard echocardiography equipment. The shockwaves are delivered in synchronization with Patient R-wave to avoid arrhythmias. The treatment is painless.

At first, the patient undergoes stress- SPECT testing to identify the ischemic areas. Following that, the same area is localized by the ultra-sound device and the shockwaves are focused to the ischemic area. Several treatments are required for optimal results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic stable angina pectoris.
* Documented myocardial segments with reversible ischemia
* AP CCS class of III-IV.
* Stable dosage of medication used to treat angina for at least 6 weeks prior to enrollment.
* Exercise tolerance time < 10 min (modified Bruce)
* Two ETT tests results (within two weeks) averaging no more than 25% of their mean
* Documented epicardial coronary artery disease not amenable to angioplasty or CABG.
* Signed an IRB approved informed consent form.
* Life expectancy of >12 months.

Exclusion Criteria:

* Intraventricular thrombus
* Malignancy in the area of treatment
* Severe COPD
* No smoking during the study procedure
* MI less <3 months prior to treatment
* Severe Valvular disease
* Child bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Total Exercise Time | 6 months

SECONDARY OUTCOMES:
Change in SPECT | 6 months
Change in AP-CCS | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Leibowitz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel